CLINICAL TRIAL: NCT04949607
Title: Traumatic Brain Injury and the Gut Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Neuro Skills (Industry)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00054911
Record Dates: First submitted 2021-06-25; First posted 2021-07-02 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Brain Injury, Chronic; Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injury, Chronic; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Subjects will be administered 1-4 grams of Inulin twice daily for 3 months.
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Traumatic Brain Injury (Experimental): Subjects aged 18-70 years with chronic traumatic brain injury receiving Inulin treatment.
  Interventions: Dietary Supplement: Inulin fructooligosaccharide
- Healthy Controls (Experimental): Healthy subjects aged 18-70 years receiving Inulin treatment.
  Interventions: Dietary Supplement: Inulin fructooligosaccharide

INTERVENTIONS:
Dietary Supplement: Inulin fructooligosaccharide — Subjects will be administered inulin at a starting dose of 1g twice daily (2g/day) and ramping up an additional 2g/day until the final dose of 4g twice daily (8g/day), which will continue on until the end of month 3 (week 12). After the month 3 study visit, inulin dosing will begin to ramp down over the next week.

SUMMARY:
The purpose of the study is to determine whether administration of a prebiotic, inulin, can improve the symptom complex associated with traumatic brain injury and whether inulin administration can alter the bacteria that live in the gut.

DETAILED DESCRIPTION:
The investigators will study subjects (aged 18-70 years) with a history of moderate/severe traumatic brain injury (n=10) and healthy controls (aged 18-70 years) (n=10). All subjects will undergo a 3-month intervention of oral inulin treatment. The traumatic brain injury subjects will be administered oral inulin twice daily for 3 months. Testing including cognitive function assessment (Repeatable Battery for the Assessment of Neuropsychological Status (RBANS), and questionnaires of fatigue, mood and quality of life and sleep will occur at month 0, 3 and 6. Blood sampling for measurement of amino acid levels, hormones, short chain fatty acids and markers of neuroinflammation will be drawn before and 90 minutes (+/- 10 minutes) after a standardized meal will occur at month 0 and month 3. In addition, fecal samples for analysis of the GI microbiome will be collected at month -1, month 0, month 1, month 2, month 3, and month 6 along with an assessment of gastrointestinal health. Traumatic brain injury subjects will be selected from residents at a long term residential rehabilitation center. Healthy control subjects will be administered oral inulin twice daily with meals for 3 months. Quality of life will be assessed by questionnaires at months 0, 3 and 6. Blood sampling for measurement of amino acid levels, hormones, short chain fatty acids and markers of neuroinflammation will be drawn before and 90 minutes (+/- 10 minutes) after a standardized meal will occur at month 0 and month 3. Fecal samples will be collected at month -1, month 0, month 3 and month 6 for analysis of the GI microbiome along with an assessment of gastrointestinal health. A member of the study team will check monthly for adverse events and overall well-being and ensure compliance and ongoing consent.

ELIGIBILITY:
Inclusion Criteria:

-Traumatic Brain Injury

Head trauma greater than two years prior manifesting in one or more of the following:

1. Loss of consciousness
2. Post-traumatic amnesia
3. Focal neurologic deficits
4. Seizures
5. Persistent symptoms of increased arousal (e.g., difficulty falling or staying asleep, anger and hypervigilance)
6. Impairment in cognitive, social, occupational, or other important areas of functioning (e.g., problems with work and relationships)

Exclusion Criteria:

* Traumatic Brain Injury

  1. Unwilling to give consent. Patients with rights managed by Legal Authorized Representative must consent to participate in addition to consent from their legal agent
  2. < 2 years post-injury
  3. Known allergy to study agent.
  4. Other medical condition or medication administration deemed exclusionary by the study investigators.

     Inclusion Criteria:
* Healthy Control

  1. Ages 18 to 70 years
  2. Works at Centre for Neuro Skills
  3. Participant is willing and able to give informed consent for participation in the study.

     Exclusion Criteria
* Healthy Control

  1. Subjects with a history of inflammatory bowel disease, Celiac disease or active diverticular disease.
  2. Known allergy to study agent.
  3. Other medical condition or medication administration deemed exclusionary by the study investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Characterization of fecal microbiome using molecular methods at baseline | Baseline
  Characterization of the fecal microbiome using a commercially available sampling kit and our lab's patented array for Polymerase Chain Reaction.
Characterization of fecal microbiome using molecular methods at month 1 | month 1
  Characterization of the fecal microbiome using a commercially available sampling kit and our lab's patented array for Polymerase Chain Reaction.
Characterization of fecal microbiome using molecular methods at month 2 | month 2
  Characterization of the fecal microbiome using a commercially available sampling kit and our lab's patented array for Polymerase Chain Reaction.
Characterization of fecal microbiome using molecular methods at month 3 | month 3
  Characterization of the fecal microbiome using a commercially available sampling kit and our lab's patented array for Polymerase Chain Reaction.
Characterization of fecal microbiome using molecular methods at month 6 | month 6
  Characterization of the fecal microbiome using a commercially available sampling kit and our lab's patented array for Polymerase Chain Reaction.

SECONDARY OUTCOMES:
Sleep Quality as measured by Pittsburgh Sleep Quality Index at baseline | Baseline (month 0)
  Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1 month-time interval. Minimum Score = 0 (better); Maximum Score = 21 (worse). Interpretation: Total < 5 associated with good sleep quality. Total > 5 associated with poor sleep quality.
Sleep Quality as measured by Pittsburgh Sleep Quality Index at month 3 | month 3
  Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1 month-time interval. Minimum Score = 0 (better); Maximum Score = 21 (worse). Interpretation: Total < 5 associated with good sleep quality. Total > 5 associated with poor sleep quality.
Sleep Quality as measured by Pittsburgh Sleep Quality Index at month 6 | month 6
  Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1 month-time interval. Minimum Score = 0 (better); Maximum Score = 21 (worse). Interpretation: Total < 5 associated with good sleep quality. Total > 5 associated with poor sleep quality.
Symptoms of Growth Hormone Deficiency measured by the questionnaire Quality of Life - Assessment of Growth Hormone Deficiency in Adults at baseline | Baseline (month 0)
  Symptoms of growth hormone deficiency will be measured using the Quality of Life - Assessment of Growth Hormone Deficiency in Adults (QoL-AGHDA). This 25-item questionnaire measures specific symptoms associated with growth hormone deficiency, with a score range of 0 to 25, with a higher score indicating worse symptoms. This assessment is completed by the Traumatic Brain Injury group only.
Symptoms of Growth Hormone Deficiency measured by the questionnaire Quality of Life - Assessment of Growth Hormone Deficiency in Adults at month 3 | month 3
  Symptoms of growth hormone deficiency will be measured using the Quality of Life - Assessment of Growth Hormone Deficiency in Adults (QoL-AGHDA). This 25-item questionnaire measures specific symptoms associated with growth hormone deficiency, with a score range of 0 to 25, with a higher score indicating worse symptoms. This assessment is completed by the Traumatic Brain Injury group only.
Symptoms of Growth Hormone Deficiency measured by the questionnaire Quality of Life - Assessment of Growth Hormone Deficiency in Adults at month 6 | month 6
  Symptoms of growth hormone deficiency will be measured using the Quality of Life - Assessment of Growth Hormone Deficiency in Adults (QoL-AGHDA). This 25-item questionnaire measures specific symptoms associated with growth hormone deficiency, with a score range of 0 to 25, with a higher score indicating worse symptoms. This assessment is completed by the Traumatic Brain Injury group only.
Depression measured by the Beck Depression Inventory-II at baseline | Baseline (month 0)
  The Beck Depression Inventory- II (BDI-II) assesses depressive symptom severity. The BDI-II is comprised of 21 individual items reflecting specific cognitive, affective, and physical symptoms of depression. Each item includes four statements that vary in the description of symptom of severity. Scores range from 0 to 3, with a score of "3" indicating a severe symptoms and a score of "0" indicating an absence of concern with that particular aspect of depressive symptomology. The total score is the sum of all endorsed statements. The maximum total score is 63. The BDI-II Manual designates the following raw score classifications depression severity: ≤13 = minimal; 14-19 = mild; 20-28 = moderate; ≥ 29 = severe.
Depression measured by the Beck Depression Inventory-II at month 3 | month 3
  The Beck Depression Inventory- II (BDI-II) assesses depressive symptom severity. The BDI-II is comprised of 21 individual items reflecting specific cognitive, affective, and physical symptoms of depression. Each item includes four statements that vary in the description of symptom of severity. Scores range from 0 to 3, with a score of "3" indicating a severe symptoms and a score of "0" indicating an absence of concern with that particular aspect of depressive symptomology. The total score is the sum of all endorsed statements. The maximum total score is 63. The BDI-II Manual designates the following raw score classifications depression severity: ≤13 = minimal; 14-19 = mild; 20-28 = moderate; ≥ 29 = severe.
Depression measured by the Beck Depression Inventory-II at month 6 | month 6
  The Beck Depression Inventory- II (BDI-II) assesses depressive symptom severity. The BDI-II is comprised of 21 individual items reflecting specific cognitive, affective, and physical symptoms of depression. Each item includes four statements that vary in the description of symptom of severity. Scores range from 0 to 3, with a score of "3" indicating a severe symptoms and a score of "0" indicating an absence of concern with that particular aspect of depressive symptomology. The total score is the sum of all endorsed statements. The maximum total score is 63. The BDI-II Manual designates the following raw score classifications depression severity: ≤13 = minimal; 14-19 = mild; 20-28 = moderate; ≥ 29 = severe.
Gastrointestinal Health measured by the Gastrointestinal Symptom Rating Scale at baseline | Baseline (month 0)
  The Gastrointestinal Symptom Rating Scale (GSRS) is a specific 15-item questionnaire. Subjects are asked to numerically score their subjective symptoms on a scale of 1-7 (1 = no discomfort at all; 7 = very severe discomfort) . The sum of the scores for all 15 items is regarded as the GSRS total score. Total scores range from 15 (best outcome) to 105 (worst outcome).
Gastrointestinal Health measured by the Gastrointestinal Symptom Rating Scale at month 1 | month 1
  The Gastrointestinal Symptom Rating Scale (GSRS) is a specific 15-item questionnaire. Subjects are asked to numerically score their subjective symptoms on a scale of 1-7 (1 = no discomfort at all; 7 = very severe discomfort) . The sum of the scores for all 15 items is regarded as the GSRS total score. Total scores range from 15 (best outcome) to 105 (worst outcome).
Gastrointestinal Health measured by the Gastrointestinal Symptom Rating Scale at month 2 | month 2
  The Gastrointestinal Symptom Rating Scale (GSRS) is a specific 15-item questionnaire. Subjects are asked to numerically score their subjective symptoms on a scale of 1-7 (1 = no discomfort at all; 7 = very severe discomfort) . The sum of the scores for all 15 items is regarded as the GSRS total score. Total scores range from 15 (best outcome) to 105 (worst outcome).
Gastrointestinal Health measured by the Gastrointestinal Symptom Rating Scale at month 3 | month 3
  The Gastrointestinal Symptom Rating Scale (GSRS) is a specific 15-item questionnaire. Subjects are asked to numerically score their subjective symptoms on a scale of 1-7 (1 = no discomfort at all; 7 = very severe discomfort) . The sum of the scores for all 15 items is regarded as the GSRS total score. Total scores range from 15 (best outcome) to 105 (worst outcome).
Gastrointestinal Health measured by the Gastrointestinal Symptom Rating Scale at month 6 | month 6
  The Gastrointestinal Symptom Rating Scale (GSRS) is a specific 15-item questionnaire. Subjects are asked to numerically score their subjective symptoms on a scale of 1-7 (1 = no discomfort at all; 7 = very severe discomfort) . The sum of the scores for all 15 items is regarded as the GSRS total score. Total scores range from 15 (best outcome) to 105 (worst outcome).
Perceptual Fatigue as measured by the Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire at baseline | Baseline (month 0)
  Perceptual fatigue and perceptual cognition will be assessed using the 20-item Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire. Each item will be measured on an individual visual analog scale of 0 - 100, where the subject will mark how true each item is for them on the line with a pencil or pen with "0" indicating "not at all" and "100" indicating "extremely". Subtests of fatigue and cognition will be measured as well as a total score. Subscores and total scores range from 0-100, with a higher score indicating worse symptoms of BIAFAC.
Perceptual Fatigue as measured by the Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire at month 3 | month 3
  Perceptual fatigue and perceptual cognition will be assessed using the 20-item Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire. Each item will be measured on an individual visual analog scale of 0 - 100, where the subject will mark how true each item is for them on the line with a pencil or pen with "0" indicating "not at all" and "100" indicating "extremely". Subtests of fatigue and cognition will be measured as well as a total score. Subscores and total scores range from 0-100, with a higher score indicating worse symptoms of BIAFAC.
Perceptual Fatigue as measured by the Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire at month 6 | month 6
  Perceptual fatigue and perceptual cognition will be assessed using the 20-item Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire. Each item will be measured on an individual visual analog scale of 0 - 100, where the subject will mark how true each item is for them on the line with a pencil or pen with "0" indicating "not at all" and "100" indicating "extremely". Subtests of fatigue and cognition will be measured as well as a total score. Subscores and total scores range from 0-100, with a higher score indicating worse symptoms of BIAFAC.
Perceptual Cognition as measured by the Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire at baseline | Baseline (month 0)
  Perceptual fatigue and perceptual cognition will be assessed using the 20-item Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire. Each item will be measured on an individual visual analog scale of 0 - 100, where the subject will mark how true each item is for them on the line with a pencil or pen with "0" indicating "not at all" and "100" indicating "extremely". Subtests of fatigue and cognition will be measured as well as a total score. Subscores and total scores range from 0-100, with a higher score indicating worse symptoms of BIAFAC.
Perceptual Cognition as measured by the Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire at month 3 | month 3
  Perceptual fatigue and perceptual cognition will be assessed using the 20-item Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire. Each item will be measured on an individual visual analog scale of 0 - 100, where the subject will mark how true each item is for them on the line with a pencil or pen with "0" indicating "not at all" and "100" indicating "extremely". Subtests of fatigue and cognition will be measured as well as a total score. Subscores and total scores range from 0-100, with a higher score indicating worse symptoms of BIAFAC.
Perceptual Cognition as measured by the Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire at month 6 | month 6
  Perceptual fatigue and perceptual cognition will be assessed using the 20-item Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire. Each item will be measured on an individual visual analog scale of 0 - 100, where the subject will mark how true each item is for them on the line with a pencil or pen with "0" indicating "not at all" and "100" indicating "extremely". Subtests of fatigue and cognition will be measured as well as a total score. Subscores and total scores range from 0-100, with a higher score indicating worse symptoms of BIAFAC.
Total BIAFAC (Brain Injury Fatigue and Altered Cognition) Score as measured by the Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire at baseline | Baseline (month 0)
  Perceptual fatigue and perceptual cognition will be assessed using the 20-item Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire. Each item will be measured on an individual visual analog scale of 0 - 100, where the subject will mark how true each item is for them on the line with a pencil or pen with "0" indicating "not at all" and "100" indicating "extremely". Subtests of fatigue and cognition will be measured as well as a total score. Subscores and total scores range from 0-100, with a higher score indicating worse symptoms of BIAFAC.
Total BIAFAC (Brain Injury Fatigue and Altered Cognition) Score as measured by the Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire at month 3 | month 3
  Perceptual fatigue and perceptual cognition will be assessed using the 20-item Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire. Each item will be measured on an individual visual analog scale of 0 - 100, where the subject will mark how true each item is for them on the line with a pencil or pen with "0" indicating "not at all" and "100" indicating "extremely". Subtests of fatigue and cognition will be measured as well as a total score. Subscores and total scores range from 0-100, with a higher score indicating worse symptoms of BIAFAC.
Total BIAFAC (Brain Injury Fatigue and Altered Cognition) Score as measured by the Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire at month 6 | month 6
  Perceptual fatigue and perceptual cognition will be assessed using the 20-item Brain Injury Fatigue and Altered Cognition (BIAFAC) Questionnaire. Each item will be measured on an individual visual analog scale of 0 - 100, where the subject will mark how true each item is for them on the line with a pencil or pen with "0" indicating "not at all" and "100" indicating "extremely". Subtests of fatigue and cognition will be measured as well as a total score. Subscores and total scores range from 0-100, with a higher score indicating worse symptoms of BIAFAC.
Cognition as assessed by the Repeatable Battery Assessment for Neuropsychological Status (RBANS) at baseline | Baseline
  The Repeatable Battery Assessment for Neuropsychological Status (RBANS) is a cognitive battery that has been utilized among Traumatic Brain Injury patients. It is comprised of 12 tests that assess five cognitive domains including immediate and delayed memory, language, visuospatial/constructional abilities, and attention. Immediate memory is assessed by two tests (list learning and story learning), visuospatial/constructional abilities is assessed by two tests (figure copy and line orientation), language is assessed by two tests (picture naming and semantic fluency), attention is two tests (digit span and coding), and delayed memory is assessed by four tests (list recall, list recognition, story recall and figure recall). RBANS raw subtests scores are converted to index standard scores. The RBANS has a mean score of 100 with a Standard Deviation of 15. Scores range from 40 to 160. Only the Traumatic Brain Injury group will undergo cognitive assessment.
Cognition as assessed by the Repeatable Battery Assessment for Neuropsychological Status (RBANS) at month 3 | month 3
  The Repeatable Battery Assessment for Neuropsychological Status (RBANS) is a cognitive battery that has been utilized among Traumatic Brain Injury patients. It is comprised of 12 tests that assess five cognitive domains including immediate and delayed memory, language, visuospatial/constructional abilities, and attention. Immediate memory is assessed by two tests (list learning and story learning), visuospatial/constructional abilities is assessed by two tests (figure copy and line orientation), language is assessed by two tests (picture naming and semantic fluency), attention is two tests (digit span and coding), and delayed memory is assessed by four tests (list recall, list recognition, story recall and figure recall). RBANS raw subtests scores are converted to index standard scores. The RBANS has a mean score of 100 with a Standard Deviation of 15. Scores range from 40 to 160. Only the Traumatic Brain Injury group will undergo cognitive assessment.
Cognition as assessed by the Repeatable Battery Assessment for Neuropsychological Status (RBANS) at month 6 | month 6
  The Repeatable Battery Assessment for Neuropsychological Status (RBANS) is a cognitive battery that has been utilized among Traumatic Brain Injury patients. It is comprised of 12 tests that assess five cognitive domains including immediate and delayed memory, language, visuospatial/constructional abilities, and attention. Immediate memory is assessed by two tests (list learning and story learning), visuospatial/constructional abilities is assessed by two tests (figure copy and line orientation), language is assessed by two tests (picture naming and semantic fluency), attention is two tests (digit span and coding), and delayed memory is assessed by four tests (list recall, list recognition, story recall and figure recall). RBANS raw subtests scores are converted to index standard scores. The RBANS has a mean score of 100 with a Standard Deviation of 15. Scores range from 40 to 160. Only the Traumatic Brain Injury group will undergo cognitive assessment.
1 methyl Histidine at baseline | Baseline (month 0)
  Amino acid 1 methyl histidine (1MHis) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
1 methyl Histidine at month 3 | month 3
  Amino acid 1 methyl histidine (1MHis) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
3 methyl Histidine at baseline | Baseline (month 0)
  Amino acid 3 methyl histidine (3MHis) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
3 methyl Histidine at month 3 | month 3
  Amino acid 3 methyl histidine (3MHis) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
L-alpha-Aminoadipic acid at baseline | Baseline (month 0)
  Amino acid L-alpha-Aminoadipic (Aad) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
L-alpha-Aminoadipic acid at month 3 | month 3
  Amino acid L-alpha-Aminoadipic (Aad) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
2-Aminobutyric Acid at baseline | Baseline (month 0)
  Amino acid 2-Aminobutyric Acid (Abu) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
2-Aminobutyric Acid at month 3 | month 3
  Amino acid 2-Aminobutyric Acid (Abu) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Alanine at baseline | Baseline (month 0)
  Amino acid Alanine (Ala) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Alanine at month 3 | month 3
  Amino acid Asparagine (Asn) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Asparagine at baseline | Baseline (month 0)
  Amino acid Asparagine (Asn) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Asparagine at baseline | month 3
  Amino acid Asparagine (Asn) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Arginine at baseline | Baseline (month 0)
  Amino acid Arginine (Arg) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Arginine at month 3 | month 3
  Amino acid Arginine (Arg) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Aspartate at baseline | Baseline (month 0)
  Amino acid Aspartate(Asp) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Aspartate at month 3 | month 3
  Amino acid Aspartate(Asp) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
D, L-beta-Aminoisobutyric acid | Baseline (month 0)
  Amino acid D, L-beta-Aminoisobutyric acid (bAid) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
D, L-beta-Aminoisobutyric acid | month 3
  Amino acid D, L-beta-Aminoisobutyric acid (bAid) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
beta-Alanine at baseline | Baseline (month 0)
  Amino acid beta-Alanine (bAla) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
beta-Alanine at month 3 | month 3
  Amino acid beta-Alanine (bAla) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
L-Carnosine | Baseline (month 0)
  Amino acid L-Carnosine (Car) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
L-Carnosine | month 3
  Amino acid L-Carnosine (Car) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Citrulline at baseline | Baseline (month 0)
  Amino acid citrulline (Cit) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Citrulline at month 3 | month 3
  Amino acid citrulline (Cit) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Cystathionine | Baseline (month 0)
  Amino acid Cystathionine (Cth) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Cystathionine | month 3
  Amino acid Cystathionine (Cth) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Cysteine at baseline | Baseline (month 0)
  Amino acid cysteine (Cys) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Cysteine at month 3 | month 3
  Amino acid cysteine (Cys) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Ethanolamine at baseline | Baseline (month 0)
  Amino acid ethanolamine (Etn) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Ethanolamine at month 3 | month 3
  Amino acid ethanolamine (Etn) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Gamma aminobutyric acid at baseline | Baseline (month 0)
  Amino acid gamma aminobutyric acid (GABA) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Gamma aminobutyric acid at month 3 | month 3
  Amino acid gamma aminobutyric acid (GABA) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Glutamine at baseline | Baseline (month 0)
  Amino acid glutamine (Gln) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Glutamine at month 3 | month 3
  Amino acid glutamine (Gln) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Glutamate at baseline | Baseline (month 0)
  Amino acid glutamate (Glu) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Glutamate at month 3 | month 3
  Amino acid glutamate (Glu) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Glycine at baseline | Baseline (month 0)
  Amino acid glycine (Gly) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Glycine at month 3 | month 3
  Amino acid glycine (Gly) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Homocysteine at baseline | Baseline (month 0)
  Amino acid homocysteine (Hcy) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Homocysteine at month 3 | month 3
  Amino acid homocysteine (Hcy) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Histidine at baseline | Baseline (month 0)
  Amino acid histidine (His) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Histidine at month 3 | month 3
  Amino acid histidine (His) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Hydroxylysine at baseline | Baseline (month 0)
  Amino acid hydroxylysine (Hyl) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Hydroxylysine at month 3 | month 3
  Amino acid hydroxylysine (Hyl) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Hydroxyproline at baseline | Baseline (month 0)
  Amino acid hydroxyproline (Hyp) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Hydroxyproline at month 3 | month 3
  Amino acid hydroxyproline (Hyp) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Isoleucine at baseline | Baseline (month 0)
  Amino acid Isoleucine (Ile) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Isoleucine at month 3 | month 3
  Amino acid Isoleucine (Ile) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Leucine at baseline | Baseline (month 0)
  Amino acid Leucine (Leu) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Leucine at month 3 | month 3
  Amino acid Leucine (Leu) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Lysine at baseline | Baseline (month 0)
  Amino acid Lysine (Lys) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Lysine at month 3 | month 3
  Amino acid Lysine (Lys) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Methionine at baseline | Baseline (month 0)
  Amino acid Methionine (Met) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Methionine at month 3 | month 3
  Amino acid Methionine (Met) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Norleucine at baseline | Baseline (month 0)
  Amino acid Norleucine (Nle) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Norleucine at month 3 | month 3
  Amino acid Norleucine (Nle) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Norvaline at baseline | Baseline (month 0)
  Amino acid Norvaline (Nva) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Norvaline at month 3 | month 3
  Amino acid Norvaline (Nva) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Ornithine at baseline | Baseline (month 0)
  Amino acid Ornithine (Orn) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Ornithine at month 3 | month 3
  Amino acid Ornithine (Orn) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
phospho-ethanolamine at baseline | Baseline (month 0)
  Amino acid phosphoethanolamine (pEtn) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
phospho-ethanolamine at month 3 | month 3
  Amino acid phosphoethanolamine (pEtn) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Phenylalanine at baseline | Baseline (month 0)
  Amino acid phenylalanine (Phe) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Phenylalanine at month 3 | month 3
  Amino acid phenylalanine (Phe) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Proline at baseline | Baseline (month 0)
  Amino acid proline (Pro) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Proline at month 3 | month 3
  Amino acid proline (Pro) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
phospho-serine at baseline | Baseline (month 0)
  Amino acid phospho-serine (pSer) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
phospho-serine at month 3 | month 3
  Amino acid phospho-serine (pSer) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Sarcosine at baseline | Baseline (month 0)
  Amino acid sarcosine (Sar) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Sarcosine at month 3 | month 3
  Amino acid sarcosine (Sar) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Serine at baseline | Baseline (month 0)
  Amino acid serine (Ser) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Serine at month 3 | month 3
  Amino acid serine (Ser) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Taurine at baseline | Baseline (month 0)
  Amino acid taurine (Tau) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Taurine at month 3 | month 3
  Amino acid taurine (Tau) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Threonine at baseline | Baseline (month 0)
  Amino acid threonine (Thr) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Threonine at month 3 | month 3
  Amino acid threonine (Thr) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Tryptophan at baseline | Baseline (month 0)
  Amino acid tryptophan (Trp) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Tryptophan at month 3 | month 3
  Amino acid tryptophan (Trp) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Tyrosine at baseline | Baseline (month 0)
  Amino acid tyrosine (Tyr) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Tyrosine at month 3 | month 3
  Amino acid tyrosine (Tyr) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Valine at baseline | Baseline (month 0)
  Amino acid valine (val) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).
Valine at month 3 | month 3
  Amino acid valine (val) will be measured in serum before and after a standardized meal. Results will be reported as change concentration in micrometers (uM).

CONTACTS AND LOCATIONS:
Overall Officials: Brent Masel, MD, Principal Investigator — Centre for Neuro Skills
Locations (1):
- Centre for Neuro Skills, Bakersfield, California, United States

IPD SHARING:
Plan to Share IPD: No